CLINICAL TRIAL: NCT03949309
Title: Pilot Study of ILIADE: Exploring Health Literacy Within Patients Hospitalized for Acute Cardiovascular Events
Brief Title: Pilot Study of ILIADE : Exploring Health Literacy Within Patients Hospitalized for Acute Cardiovascular Events
Acronym: P-ILIADE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0207; 2019-A00799-48 (Other: ID-RCB)
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Acute Myocardial Infarction; Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible patients: All eligible patients discharged from hospital for Acute Myocardial Infarction (AMI) or acute decompensation of Chronic Heart Failure (CHF)
  Interventions: Other: Exploring health literacy levels and patients' informal needs or individual relationship between caregivers and patients.

INTERVENTIONS:
Other: Exploring health literacy levels and patients' informal needs or individual relationship between caregivers and patients. — It is a cross-sectional study coupled with a qualitative ancillary study conducted within patients hospitalized for one of the two acute cardiovascular diseases (acute coronary syndrome or acute heart failure). All patients hospitalized at Hospices Civils de Lyon for one of these two diseases and whom are going back home will be enrolled. Few patients will be interviewed during the follow-up visit at 1-month post hospitalisation. Caregivers from cardiology units will also be interviewed.

SUMMARY:
Health literacy (HL) is the ability to access, understand, evaluate and apply information in order to communicate with health professionals and understand health instructions but also, promote, maintain and improve health throughout life. Health literacy is known as a health determinant. An association has been shown between low health literacy and low health outcomes such as increased number of unscheduled hospitalization or emergency visits, low medication adherence and poor health status.

These have been particularly demonstrated with cardiovascular diseases, which combine risk factors (emergency hospitalization, reduction in the length of hospital stays, and complex secondary preventive drug treatments). Despite many scientific international literature about health literacy and health outcomes, no information is available in France on the prevalence of low health literacy level of patients, notably cardiovascular patients. The investigating team's hypothesis is that knowing the prevalence of low HL levels in cardiovascular patients would help to better tailored a communication intervention dedicated to the needs of these low-HL patients with the final aim of increasing their adhesion to preventive drugs and behavioural recommendations.

The first aim of the present study is to estimate the prevalence of low HL level among patients discharged after acute myocardial infarction or acute decompensation of chronic heart failure. Secondary aims are to assess factors associated with the level of HL and identify barriers and facilitators of low HL patients to understand medical information on their disease. The results of this study will guide the design of the intervention of an interventional study on HL of cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

- Patient

* Age greater than or equal to 18 years
* Hospitalization for Acute coronary syndrome (ACS) (myocardial infarction with or without ST segment elevation) or acute attack of heart failure (systolic or diastolic)
* Able to communicate in French and/or helping to communicate in French
* Return home after hospitalization

Health professional

* Voluntary and available for the entire interview
* Having participated in the management of the patient screened on the day of the consultation
* Cardiologist, intern or emergency department nurse
* Attached to the participating service

Exclusion Criteria:

- Patient

* Short-term vital prognosis
* Severe dementia
* Inability to manage drug treatment alone
* Institutionalization at the end of hospitalization

Health professional

* Health professional working in the department only one or two days a week
* Health professional who is not specialized in diseases of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized for Acute myocardial infarction (AMI) and acute decompensation of chronic heart failure (CHF) will be screened for one month in the cardiology departments of the Louis Pradel Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Brief Health Literacy Screening (BHLS) of patients hospitalized for a cardiovascular disease. | Day 1
  Health literacy will be measured thanks to the questionnaire Brief Health Literacy Screening (BHLS). This questionnaire is composed of 3 questions and is known to screen quickly patient health literacy. The 3 responses are summed to generate a score between 3 and 15, where higher scores indicated higher health literacy. Low health literacy is defined as Brief Health Literacy Screen less than or equal to a score of 9.

SECONDARY OUTCOMES:
Health Literacy Questionnaire (HLQ) | Day 1
  The HLQ explores more dimensions of health literacy such as social support relationship with caregivers, health information evaluation or ability to engage with caregivers. It consists of 44 items. Participants are asked to rate "How strongly do you disagree or agree with the following statements?". The options provided were: 'strongly disagree', 'disagree', 'agree' and 'strongly agree', which were scored from 1 to 4, respectively. In 2nd part of the HLQ, participants were asked "How easy or difficult are the following tasks for you to do now?" The options for these scales were 'cannot do', 'very difficult', 'quite difficult', 'quite easy' and 'very easy', which were scored from 1 to 5, respectively. The higher the score the higher the health literacy of a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie SCHOTT, PhD, Principal Investigator — Hospices Civils de Lyon; Julie HAESEBAERT, MD, Study Chair — Hospices Civils de Lyon
Locations (1):
- Groupement Hospitalier Est, Bron, France

REFERENCES:
- [Derived] Perrin A, Damiolini E, Schott AM, Zermati J, Bravant E, Delahaye F, Dima AL, Haesebaert J. Considering health literacy in cardiovascular disease management: a qualitative study on healthcare professionals' and patients' perspectives. BMC Health Serv Res. 2022 Sep 5;22(1):1121. doi: 10.1186/s12913-022-08455-8. PMID 36064395